CLINICAL TRIAL: NCT05200650
Title: A Single Arm, Prospective, Open Label, Multi Center, Phase Ib Study to Evaluate the Safety, Tolerability and Initial Efficacy of a Single Intra-tumoral Injection of IntraGel's Polymer-based Cisplatin-loaded Gel (TumoCure) in Subjects With Progressive or Radio-resistant Primary Head and Neck Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IntraGel Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLPR-001
Record Dates: First submitted 2021-12-30; First posted 2022-01-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TumoCure Treatment (Experimental): Subjects will be treated with a single intra-tumor injection of TumoCure, containing the polymeric delivery system and the Cisplatin hemotherapy agent at a dose of 100mg.
  Interventions: Combination Product: TumoCure

INTERVENTIONS:
Combination Product: TumoCure — TumoCure is a polymer-based gel, loaded with Cisplatin in a dose of 100mg (10% w/w), injected to head and neck tumors locally in a single injection.

SUMMARY:
IntraGel's polymer-based Cisplatin loaded Gel (TumoCure) is a single injectable compound, aimed at localized chemotherapy treatment. The treatment is offered to patients who currently have no other available treatment options, either due to inefficacy, intolerability or inapplicability of standard treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18-80 years.
2. Subjects who are willing to comply with study procedures.
3. Subjects who are mentally and cognitively capable and who are capable of understanding and signing the informed consent.
4. Subjects with a known diagnosis of primary head and neck cancer, with or without metastases.
5. Subjects with a progressing or radio-resistant disease, who are unable, unwilling or do not tolerate currently available treatments.
6. Subjects with a measurable tumor by either ultrasound, MRI or CT.
7. Subjects with ECOG performance status of 0 -2.

Exclusion Criteria:

1. Subjects with life expectancy of less than 3 months.
2. Pregnant or breastfeeding women.
3. Known COPD or other chronic pulmonary or respiratory disease, with PFT's indicating a FEV<50% predicted for age.
4. Known reduced renal function, defined S-Creatinine ≥ 1.5xULN or Creatinine clearance < 40 ml/min, calculated by using the Cockroft and Gault formula.
5. Reduced hepatic function, defined as ASAT, ALAT, bilirubin > 1.5xULN and PK-INR > 1.5, or a known medical history of liver cirrhosis or portal hypertension.
6. Blood leukocytes count <1.5 *103/microl or platelets <75 *103/microl.
7. Subject who was treated with systemic chemotherapy during the 4 weeks preceding screening.
8. Participation in any other clinical trial that included an investigational device or medicinal product.
9. Any other condition that according to the discretion of the primary investigator precludes the subject from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Adverse Events | 90 days
  Cumulative rate of treatment - related serious adverse events (SAEs) throughout the follow up period (90 days)

SECONDARY OUTCOMES:
Change in Tumor Size (Efficacy) | 90 days
  change in tumor size from baseline to the end of the follow up period (90 days) according to the RECIST methodology, as determined by MRI/CT imaging

OTHER OUTCOMES:
Overall Survival | 90 days
  Overall survival (OS) throughout the follow up period (90 days)
Subject Quality of Life | 90 days
  Subject Quality of Life (QoL), as determined by the change in EORTC-QLQ30 (European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire - 30) total score (ranging from 30-120, the lower the result, the better quality of life the subject reports) from baseline to end of follow up period.
Subject Quality of Life | 90 days
  EORTC-QLQ HNC43 (European Organization for Research and Treatment of Cancer - Quality of Life Head and Neck Questionnaire 43) questionnaire total score (ranging from 43-172, the lower the result the better quality of life the subject reports) from baseline to end of follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Aharon Popovizer, MD, Principal Investigator — Head of Head and Neck Surgery Department
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be shared